CLINICAL TRIAL: NCT06185205
Title: Accelerated Super-Hypofractionated Breast Brachytherapy - ASHBY Trial
Brief Title: ASHBY: Accelerated Super-Hypofractionated Breast Brachytherapy
Acronym: ASHBY
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-22-19248; HM20027787 (Other: Virginia Commonwealth University)
Record Dates: First submitted 2023-12-14; First posted 2023-12-29 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Ductal Carcinoma in situ (DCIS); Irradiation
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Accelerated Partial Breast Irradiation (APBI) (Experimental): 7.5 gray (Gy) × 3 fractions via multicatheter brachytherapy
  Interventions: Drug: Accelerated partial breast irradiation

INTERVENTIONS:
Drug: Accelerated partial breast irradiation — High Dose Rate treatment delivery

SUMMARY:
The purpose of this study is to compare any good and bad effects of giving radiation treatment for breast cancer in 3 treatments over about 2 days.

DETAILED DESCRIPTION:
This phase 2, single-arm prospective study has been designed to determine the safety of delivering accelerated partial breast irradiation (APBI) with a multicatheter interstitial implant in a short course over 1.5 days

ELIGIBILITY:
Inclusion Criteria:

* Female
* New diagnosis of ductal carcinoma in situ (DCIS) and/or invasive breast carcinoma per histologic evaluation
* Age 45-79 at diagnosis
* Previous lumpectomy with surgical margins histologically free of invasive tumor and DCIS as determined by the pathologist.
* T stage of Tis, T1, or T2.
* T2 tumors must be ≤3 cm in maximum diameter
* If the tumor is human epidermal growth factor receptor 2 (HER2)-positive, the patient must receive HER2-directed therapy.
* For patients with invasive breast cancer, an axillary staging procedure must be performed (either sentinel node biopsy alone or axillary dissection [with a minimum of 6 axillary nodes removed]) and the axillary node[s] must be pathologically negative.
* Note: N0(i+) is not an exclusion criterion.
* Note: Patients meeting all of the following criteria are not required to undergo the axillary staging procedure:

  * ≥70 years of age
  * estrogen receptor, Her2 = human epidermal growth factor receptor 2, PR = progesterone receptor negative (ER+PR+HER2-)
  * G1-2
  * Tumor ≤2 cm in size
  * Agrees to comply with aromatase inhibitor recommendation
* Ability to understand and the willingness to sign a written informed consent document in English

Exclusion Criteria:

* Pregnant or breastfeeding
* Active collagen-vascular disease
* Paget's disease of the breast
* History of DCIS or invasive breast cancer prior to the current diagnosis
* Prior breast or thoracic radiation therapy (RT) for any condition
* Multicentric carcinoma (DCIS or invasive)
* Synchronous bilateral invasive or non-invasive breast cancer
* Surgical margins that cannot be microscopically assessed or that are positive
* Excision cavity that cannot be clearly delineated per the treating investigator
* Any of the dosimetric treatment criteria defined in Section 6.1 have not been met. Patients who become ineligible due to inability to meet dosimetric criteria should not receive treatment as - defined in this protocol and will come off the study. Any subsequent adjuvant radiation will be delivered at the discretion of the treating physician
* Medical, psychological, or social condition that, in the opinion of the investigator, may increase the patient's risk or limit the patient's adherence with study requirements

Ages: 45 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2031-01-31 (Estimated); Study Completion 2033-01-31 (Estimated)

PRIMARY OUTCOMES:
Assess the toxicity (at 1 and 3 years) of a 1.5-day APBI treatment course | 1 year, and 5 years following irradiation
  Determine the incidence of accelerated partial breast irradiation (APBI) related toxicities, adverse events, of interest occurring at grade ≥3 within 1 year and 3 years after APBI. The APBI-related toxicities specified in Section 10.1 will be explicitly evaluated at all follow-up appointments. All APBI-related toxicities of interest will be captured, regardless of grade, beginning with the start of study treatment and continuing until the patient is off study utilizing study-specific grading criteria in place of Common Terminology Criteria for Adverse Events (CTCAE) v5.0.

SECONDARY OUTCOMES:
Assess the rate of excellent or good cosmesis at baseline, 1, 3, and 5 years after a 1.5-day course of APBI utilizing the Breast Cancer Treatment Outcome Scale. | Baseline, one year, three years, and five years following irradiation
  Cosmesis will be assessed utilizing the Breast Cancer Treatment Outcome Scale (BCTOS-12), a self-report instrument that evaluated the aesthetic outcome after breast conserving surgery (BCS). the Aesthetic Status, is composed of eight items referring to the breast. the new Aesthetic Status comprises eight items: (1) "breast shape", (2) "breast texture", (3) "nipple appearance", (4) "breast tenderness", (5) "scar tissue", (6) "breast swelling", (7) "fit of bra", and (8) "breast sensitivity".
  Patients are instructed to rate each item of the BCTOS questionnaire on a four-point rating scale evaluating the differences between the treated and untreated breast (1 = no difference to 4 = large difference). The score for each subscale is calculated as the mean of its items, with the score ranging from 1.00 to 4.00. A higher score reflects a poorer status.
Assess the rate of excellent or good cosmesis at baseline, 1, 3, and 5 years after a 1.5-day course of APBI utilizing the Breast Cancer Treatment Outcome Scale. | Baseline, one year, three years, and five years following irradiation
  Cosmesis will be assessed utilizing the Breast Cancer Treatment Outcome Scale (BCTOS-12), a self-report instrument that evaluated the functional outcome after breast conserving surgery (BCS). The questionnaire comprises 12 items and assesses various aspects of patients' subjective perception of the surgical result. The new Functional Status comprises four items: (1) "arm heaviness", (2) "shoulder discomfort", (3) "arm discomfort", (4) "arm swelling". Patients are instructed to rate each item of the BCTOS questionnaire on a four-point rating scale evaluating the differences between the treated and untreated breast
  (1 = no difference to 4 = large difference). The score for each subscale is calculated as the mean of its items, with the score ranging from 1.00 to 4.00. A higher score reflects a poorer status.
Assess the rate of excellent or good cosmesis at baseline, 1, 3, and 5 years after a 1.5-day course of APBI utilizing the BREAST-Q©. | Baseline, one year, three years, and five years following irradiation
  The radiation-specific module of this patient-reported outcome measure evaluates patient satisfaction with the cosmetic effects of radiation by utilizing the BREAST-Q© (intellectual property of Drs Andrea Pusic, Anne Klassen and Stefan Cano. The BREAST-Q© is owned by Memorial Sloan Kettering Cancer Center and The University of British Columbia (Copyright ©2012, Memorial Sloan Kettering Cancer Center and The University of British Columbia). There is no overall or total BREAST-Q© score, only scores for each independent scale. All BREAST-Q© scales are transformed into scores that range from 0-100. The scores are computed by adding the response items together and then converting the raw sum scale score to a score from 0-100. For all BREAST-Q© scales, a higher score means greater satisfaction or better QOL.
Assess the rate of excellent or good cosmesis at baseline, 1, 3, and 5 years after a 1.5-day course of APBI utilizing the Harvard Cosmesis Scale | Baseline, one year, three years, and five years following irradiation
  This physician-rated form will be used by the treating surgeon or radiation oncologist to score cosmesis at baseline and annually for 5 years, where Excellent= treated breast looks essentially the same as the contralateral breast as it relates to radiation effects. This includes patients with grade 1 punctate scarring. Good= minimal but identifiable radiation effects of the treated breast. This includes patients with grade 2 punctate scarring.
  Fair= significant radiation effects readily observable. Poor= severe sequelae of breast tissue secondary to radiation effect
Determine the 3- and 5-year actuarial local control rate of breast cancer when treated with a 1.5-day course of APBI. | up to three and five years after irradiation
  The number of participants that achieve complete responses, partial response, or relapse. Disease control will be assessed by physical examination and mammography.
Assess cumulative treatment-related breast toxicities for up to 5 years after a 1.5-day course of APBI | up to five years after irradiation
  The number of participants that have a reportable adverse event (AE) per protocol criteria.
Conduct detailed evaluation of the severity of punctate scarring at 5 weeks, 6 months, and yearly through 5 years after a 1.5-day course of APBI | 5 weeks, 6 months, and yearly through 5 years following irradiation
  Incidence and grade of punctate scarring. Punctate scarring, defined as scarring from catheter sites, is assigned according to the following grading criteria (Table 5):
  * No toxicity: not clearly visible from 3 feet away
  * Grade 1a: clearly visible from 3 feet away and no palpable scars
  * Grade 1b: clearly visible from 3 feet away and palpable scars at <25% of catheter sites) OR clearly visible at 3-10 feet and no palpable scar tissue
  * Grade 1c: clearly visible from ≥10 feet away and no palpable scars OR clearly visible at <10 feet and palpable scars at <25% of catheter sites)
  * Grade 2: prominent (ie, visible at ≥10 feet away) and palpable scar tissue
Assess rates of skin changes after a 1.5-day course of APBI in African American and non-African American patients. | 5 weeks, 6 months, and yearly through 5 years following irradiation
  Incidence of skin changes after APBI in African American and non-African American patients.

CONTACTS AND LOCATIONS:
Overall Officials: Bridget Quinn, MD, Ph.D, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No